CLINICAL TRIAL: NCT04153110
Title: Cerebello-Spinal tDCS as Rehabilitative Intervention in Neurodegenerative Ataxias: a Randomized, Double-blind, Sham-controlled Trial Followed by an Open-label Phase
Brief Title: Cerebello-Spinal tDCS as Rehabilitative Intervention in Neurodegenerative Ataxia
Acronym: SCA02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP3244
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Ataxia; Spinocerebellar Ataxias; Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia 3; Multiple System Atrophy; Ataxia With Oculomotor Apraxia; CANVAS
Keywords: Transcranial direct current stimulation; Transcranial magnetic stimulation; Spinocerebellar ataxia; Cerebellar ataxia
MeSH Terms: conditions — Ataxia; Spinocerebellar Ataxias; Machado-Joseph Disease; Multiple System Atrophy; Spinocerebellar ataxia, autosomal recessive 1; Cerebellar Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS - Real tDCS (Experimental): 10 sessions of anodal cerebellar and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks) followed by an open-label 10 sessions of anodal cerebellar and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks)
  Interventions: Device: Anodal cerebellar and cathodal spinal tDCS
- Sham tDCS - Real tDCS (Sham Comparator): 10 sessions of sham cerebellar and sham spinal transcranial direct current stimulation (5 days/week for 2 weeks) followed by an open-label 10 sessions of anodal cerebellar and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks).
  Interventions: Device: Anodal cerebellar and cathodal spinal tDCS; Device: Sham cerebellar and sham spinal tDCS

INTERVENTIONS:
Device: Anodal cerebellar and cathodal spinal tDCS — 10 sessions of anodal cerebellar and cathodal spinal transcranial direct current stimulation (5 days/week for 2 weeks)
Device: Sham cerebellar and sham spinal tDCS — 10 sessions of sham cerebellar and sham spinal transcranial direct current stimulation (5 days/week for 2 weeks)
  Arms: Sham tDCS - Real tDCS

SUMMARY:
Neurodegenerative cerebellar ataxias represent a group of disabling disorders which currently lack effective therapies. Cerebellar transcranial direct current stimulation (tDCS) is a non-invasive technique, which has been demonstrated to modulate cerebellar excitability and improve symptoms in patients with cerebellar ataxias. In this randomized, double-blind, sham-controlled study followed by an open-label phase, the investigators will evaluate whether a repetition of two-weeks' treatment with cerebellar anodal tDCS and spinal cathodal tDCS, after a three months interval, may further outlast clinical improvement in patients with neurodegenerative cerebellar ataxia and can modulate cerebello-motor connectivity, at short and long term.

DETAILED DESCRIPTION:
Neurodegenerative cerebellar ataxias represent a heterogeneous group of disabling disorders in which progressive ataxia of gait, limb dysmetria, oculomotor deficits, dysarthria and kinetic tremor are the prominent clinical manifestations. Both the hereditary and sporadic forms usually present in young adulthood, and are characterized by atrophy of cerebellar or brainstem structures. Currently, cerebellar ataxia lack effective disease-modifying therapies.

Cerebellar transcranial direct current stimulation (tDCS) is a non-invasive technique, which has been demonstrated to modulate cerebellar excitability and improve symptoms in patients with cerebellar ataxias. The present randomized, double-blind, sham-controlled study followed by an open-label phase will investigate a repetition of two-weeks' treatment with cerebellar anodal tDCS and spinal cathodal tDCS, after a three months interval, may further outlast clinical improvement in patients with neurodegenerative cerebellar ataxia and can modulate cerebello-motor connectivity, at short and long term. In addition the investigators will evaluate if tDCS intervention might improve cerebellar cognitive-affective syndrome in patients with ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cerebellar syndrome and quantifiable cerebellar atrophy

Exclusion Criteria:

* Severe head trauma in the past
* History of seizures
* History of ischemic stroke or hemorrhage
* Pacemaker
* Metal implants in the head/neck region
* Severe comorbidity
* Intake of illegal drugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change in the International Cooperative Ataxia Rating Scale (ICARS) Score From Baseline | Baseline - 2 weeks
  International Cooperative Ataxia Rating Scale (ICARS): semi-quantitative 100-point scale, yielding a total score of 0 (no ataxia) to 100 (most severe ataxia).
Change in the Scale for the Assessment and Rating of Ataxia (SARA) Score From Baseline | Baseline - 2 weeks
  Scale for the Assessment and Rating of Ataxia (SARA): 8-item performance based scale, yielding a total score of 0 (no ataxia) to 40 (most severe ataxia).
Change in the Cerebellar cognitive affective syndrome (CCAS) Scale From Baseline | Baseline - 2 weeks
  CCAS/Schmahmann syndrome scale: 120 point scale, yielding a total score of 0 (most severe cognitive impairment) to 120 (no cognitive impairment).

SECONDARY OUTCOMES:
Change in the International Cooperative Ataxia Rating Scale (ICARS) Score From Baseline | Baseline - 2 weeks - 3 month - 6 months - 9 months
  International Cooperative Ataxia Rating Scale (ICARS): semi-quantitative 100-point scale, yielding a total score of 0 (no ataxia) to 100 (most severe ataxia).
Change in the Scale for the Assessment and Rating of Ataxia (SARA) Score From Baseline | Baseline - 2 weeks - 3 month - 6 months - 9 months
  Scale for the Assessment and Rating of Ataxia (SARA): 8-item performance based scale, yielding a total score of 0 (no ataxia) to 40 (most severe ataxia).
Change in the Cerebellar cognitive affective syndrome (CCAS) Scale From Baseline | Baseline - 2 weeks - 3 month - 6 months - 9 months
  CCAS/Schmahmann syndrome scale: 120 point scale, yielding a total score of 0 (most severe cognitive impairment) to 120 (no cognitive impairment).
Change in Cerebellar Brain Inhibition (CBI) Measurements From Baseline | Baseline - 2 weeks - 3 month - 6 months - 9 months
  Cerebellar brain inhibition (CBI) is expressed as motor evoked potential amplitude (average of 10 recordings). Lower values reflect higher inhibition and thus reduced impairment.
Change in the Short-Form Health Survey 36 (SF36) Score From Baseline | Baseline - 2 weeks - 3 month - 6 months - 9 months
  The Italian version of the Short-Form Health Survey 36 (SF-36): consists of 36 scaled score, yielding a total score of 0 (more disability) to 100 (less disability).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — Azienda Ospedaliera Spedali Civili, Brescia; Alberto Benussi, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- AO Spedali Civili, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benussi A, Dell'Era V, Cantoni V, Bonetta E, Grasso R, Manenti R, Cotelli M, Padovani A, Borroni B. Cerebello-spinal tDCS in ataxia: A randomized, double-blind, sham-controlled, crossover trial. Neurology. 2018 Sep 18;91(12):e1090-e1101. doi: 10.1212/WNL.0000000000006210. Epub 2018 Aug 22. PMID 30135258
- [Background] Benussi A, Dell'Era V, Cotelli MS, Turla M, Casali C, Padovani A, Borroni B. Long term clinical and neurophysiological effects of cerebellar transcranial direct current stimulation in patients with neurodegenerative ataxia. Brain Stimul. 2017 Mar-Apr;10(2):242-250. doi: 10.1016/j.brs.2016.11.001. Epub 2016 Nov 3. PMID 27838276
- [Background] Benussi A, Koch G, Cotelli M, Padovani A, Borroni B. Cerebellar transcranial direct current stimulation in patients with ataxia: A double-blind, randomized, sham-controlled study. Mov Disord. 2015 Oct;30(12):1701-5. doi: 10.1002/mds.26356. Epub 2015 Aug 14. PMID 26274840
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Miranda PC, Salvador R, Wenger C, Fernandes SR. Computational models of non-invasive brain and spinal cord stimulation. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:6457-6460. doi: 10.1109/EMBC.2016.7592207. PMID 28269725
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Fiocchi S, Ravazzani P, Priori A, Parazzini M. Cerebellar and Spinal Direct Current Stimulation in Children: Computational Modeling of the Induced Electric Field. Front Hum Neurosci. 2016 Oct 17;10:522. doi: 10.3389/fnhum.2016.00522. eCollection 2016. PMID 27799905
- [Background] van Dun K, Bodranghien F, Manto M, Marien P. Targeting the Cerebellum by Noninvasive Neurostimulation: a Review. Cerebellum. 2017 Jun;16(3):695-741. doi: 10.1007/s12311-016-0840-7. PMID 28032321

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT04153110/Prot_SAP_001.pdf